CLINICAL TRIAL: NCT05162365
Title: A Safety, Tolerability, and Efficacy Study of IBI314 in Ambulatory Patients With COVID-19
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The company decision that terminated the further develop of the molecule and had notified FDA about the termination as well.
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI314A201
Record Dates: First submitted 2021-12-12; First posted 2021-12-17 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — P5-22 and P14-44 drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IBI314 (Experimental): a cocktail of two SARS-CoV-2 S protein IgG1 antibodies, IBI314-A and IBI314-B, in a 1:1 [w/w] ratio
  Interventions: Biological: IBI314
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IBI314 — Low/medium/high dose, intravenously, once, on Day 1
  Arms: IBI314
Other: Placebo — Placebo, intravenously, once, on Day 1
  Arms: Placebo

SUMMARY:
This is a dose-finding, inferentially seamless Phase 1/2 study evaluating the safety, tolerability and efficacy of IBI314 in Ambulatory Patients with COVID-19.

DETAILED DESCRIPTION:
Phase 1 is a randomized, double-blind, placebo-controlled, single ascending dose study in up to 32 ambulatory adult patients with COVID-19. This phase of the study is designed to assess the safety, tolerability, PK, and PD of IBI314 administered as a single IV infusion. Phase 2 is a randomized, double-blind, placebo-controlled expansion study in approximately 208 ambulatory adult patients with COVID-19. This phase of the study is designed to assess the efficacy and safety of IBI314, administered by single IV infusion at dose levels that meet none of the termination criteria for dose escalation in Phase 1 of the study.

ELIGIBILITY:
Main Inclusion Criteria:

1. First onset of COVID-19 symptoms <7 days at randomization, symptoms such as fever and/or chills, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, and diarrhea.
2. Have a positive SARS-CoV-2 Reverse Transcription-Polymerase Chain Reaction (RT-PCR) test using an appropriate sample such as nasopharyngeal (NP), nasal, oropharyngeal, or saliva within 72 hours prior to randomization. A historical record of a positive result from a test conducted ≤72 hours prior to randomization is acceptable.
3. Male or female patients ≥18 years of age at the time of signing informed consent.
4. Agree to use an adequate method of contraception throughout the study period and for 90 days after the dose of study drug is administered.
5. Women of childbearing potential (WOCBP) must have a negative urinary pregnancy test at screening.

Main Exclusion Criteria:

1. according to protocol v3.0, Note: Patients with mild-to-moderate disease who are placed in a facility where required by local guidelines can be enrolled.
2. Have oxygen saturation (SpO2) ≤93 % on room air at sea level or a ratio of arterial oxygen partial pressure (PaO2 in millimeters of mercury) to fractional inspired oxygen (FiO2) <300, respiratory rate ≥30 per minute, heart rate ≥125 per minute.
3. Have evidence of multi-organ dysfunction/failure.
4. Systolic blood pressure <90 mmHg, diastolic blood pressure <60 mmHg, or requiring vasopressors.
5. Require or anticipated impending need for endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula noninvasive positive pressure ventilation, extracorporeal membrane oxygenation (ECMO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Number of treatment related AEs | 29 days after the last participant is randomized
  Any AEs and SAEs occurring during the study
Virologic efficacy Evaluation | 7 days after the last participant is randomized
  Time-weighted average change in viral shedding from baseline through Day 7 as measured by RT-qPCR in NP swab samples.

SECONDARY OUTCOMES:
maximum concentration (Cmax) | 29 days after the last participant is randomized
  PK parameters to be evaluated for IBI314 including maximum concentration (Cmax) will be determined when appropriate.
area under the concentration-time curve (AUC) | 29 days after the last participant is randomized
  PK parameters to be evaluated for IBI314 including area under the concentration-time curve (AUC) will be determined when appropriate.
half-life (t1/2) | 29 days after the last participant is randomized
  PK parameters to be evaluated for IBI314 including half-life (t1/2) will be determined when appropriate.
  * Time to alleviation of symptoms (going to mild or absent);
  * Proportion of patients admitted to a hospital and emergency room visit due to COVID-19 by Day 29;
  * Proportion of patients with all-cause mortality by Day 29.
clearance (CL) | 29 days after the last participant is randomized
  PK parameters to be evaluated for IBI314 including clearance (CL) will be determined when appropriate.
  * Change from baseline in viral shedding on Day 7, 11, 22;
  * Time-weighted average change in viral shedding from baseline through D11 as measured by RT-qPCR in NP swab samples;
  * Time-weighted average change in viral shedding from baseline through D22 as measured by RT-qPCR in NP swab samples.
volume of distribution (V) | 29 days after the last participant is randomized
  PK parameters to be evaluated for IBI314 including volume of distribution (V) will be determined when appropriate.
The incidence of anti-IBI314 antibody (ADA) and neutralizing antibody (NAb) in serum before and after study drug administration | 29 days after the last participant is randomized
  Each patient will be tested for anti-drug (IBI314) antibody (ADA), and ADA-positive serum samples will continue to be tested for neutralizing antibodies (NAb).
Proportion of patients with at least one COVID-19 related medically attended visits by Day 29 | 29 days after the last participant is randomized
  This is a clinical efficacy outcome measure.
Time to alleviation of symptoms (going to mild or absent) | 29 days after the last participant is randomized
  This is a clinical efficacy outcome measure.
Proportion of patients admitted to a hospital and emergency room visit due to COVID-19 by Day 29 | 29 days after the last participant is randomized
  This is a clinical efficacy outcome measure.
Proportion of patients with all-cause mortality by Day 29 | 29 days after the last participant is randomized
  This is a clinical efficacy outcome measure.
Time to negative RT-qPCR in NP swab samples with no subsequent positive RT-qPCR | 29 days after the last participant is randomized
  This is a virologic efficacy outcome measure.
Change from baseline in viral shedding on Day 7, 11, 22 | 29 days after the last participant is randomized
  This is a virologic efficacy outcome measure.
Time-weighted average change in viral shedding from baseline through D11 as measured by RT-qPCR in NP swab samples | 29 days after the last participant is randomized
  This is a virologic efficacy outcome measure.
Time-weighted average change in viral shedding from baseline through D22 as measured by RT-qPCR in NP swab samples. | 29 days after the last participant is randomized
  This is a virologic efficacy outcome measure.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Sobh, Anaheim, California
  - Long Beach Clinical Trials, LLC, Long Beach, California
  - Acclaim Clinical Research, San Diego, California
  - Herco Research Center, Inc., Coral Gables, Florida
  - Midland Florida Clinical Research Center - Inf. Disease/Infectiology, DeLand, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Sweet Hope Research Specialty, Inc, Hialeah, Florida
  - Prestige Clinical Research Center Inc, Miami, Florida
  - Cordova Research Institute, LLC, Miami, Florida
  - Clinical Trials of Florida, LLC, Miami, Florida
  - The Clinical Research Institute LLC, Miami Gardens, Florida
  - Pembroke Clinical Trials, Pembroke Pines, Florida
  - Luminous Clinical Research LLC - South Florida Urgent Care - Infectious Diseases, Pembroke Pines, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - Excel Clinical Research - Internal Medicine, Las Vegas, Nevada
  - Temple University Health System - Temple Lung Center, Philadelphia, Pennsylvania
  - Zenos Clinical Research, Dallas, Texas
  - Epic Clinical Research, Lewisville, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Y, Lin Z, Guo X, Zhang F, Wang Y, Zhang Z, Chen J, Liu L, Zhu M, Li Y, Ni M, Zhen Z, Wu Z, Ling X, Zhou S, Xi Y, Yu Y, Liang W, Zhao J, Li L, He J, Sang L. Development of broadly neutralizing antibodies against Omicron variants from existing neutralizing antibodies in clinical trials. Virol J. 2025 Nov 4;22(1):358. doi: 10.1186/s12985-025-02964-8. PMID 41188882